CLINICAL TRIAL: NCT01227603
Title: Single Dose Study to Compare the Pharmacokinetics as Well as Safety and Tolerability of a Novel Fixed Dose Combination of Nifedipine GITS and Candesartan, the Loose Combination of Both and the Single Components Alone and to Investigate the Bioequivalence Between the Fixed Dose and the Loose Combination in Healthy Male Volunteers Under Fasting Conditions in an Open Label, Randomized, 4-way-crossover Design
Brief Title: Single Dose Bioequivalence Study Comparing Nifedipine/Candesartan FDC (Fixed Dose Combination) With Loose Combination of Nifedipine GITS (Gastro-intestinal Therapeutic System) Plus Candesartan and Single Components Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14027; 2010-021966-31 (EudraCT Number)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension, Essential
Keywords: Bioequivalence; Nifedipine; Candesartan; FDC
MeSH Terms: conditions — Essential Hypertension | interventions — Nifedipine; candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nifedipine-candesartan FDC (Experimental): Each subject received single fixed dose combination of 60 mg nifedipine and 32 mg candesartan orally.
  Interventions: Drug: Nifedipine-candesartan FDC (BAY 98-7106)
- Nifedipine and candesartan (Active Comparator): Each subject received one dose of nifedipine GITS 60 mg and candesartan 32 mg (2 x 16 mg tablet) as loose combination, orally.
  Interventions: Drug: Nifedipine GITS (Adalat LA, BAYA1040); Drug: Candesartan (Atacand)
- Nifedipine (Active Comparator): Each subject received one dose of nifedipine GITS 60 mg orally.
  Interventions: Drug: Nifedipine GITS (Adalat LA, BAYA1040)
- Candesartan (Active Comparator): Each subject received one dose of candesartan 32 mg (2 x 16 mg tablet), orally.
  Interventions: Drug: Candesartan (Atacand)

INTERVENTIONS:
Drug: Nifedipine-candesartan FDC (BAY 98-7106) — Single dose of 1 FDC tablet consisting of 60 mg nifedipine GITS and 32 mg candesartan
  Arms: Nifedipine-candesartan FDC
Drug: Nifedipine GITS (Adalat LA, BAYA1040) — Single oral dose of 1 tablet of nifedipine GITS 60 mg
  Arms: Nifedipine; Nifedipine and candesartan
Drug: Candesartan (Atacand) — Single oral dose of 32 mg (2 x 16 mg tablet) candesartan
  Arms: Candesartan; Nifedipine and candesartan

SUMMARY:
Randomized, open label, single dose, 4-way crossover study to investigate the bioequivalence of a new fixed dose combination tablet of nifedipine GITS and candesartan with the corresponding loose combination and to compare it with the individual drugs

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening / examination visit
* Ethnicity: Caucasian
* Body mass index (BMI): >/=18 and </=29,9 kg/m²

Exclusion Criteria:

* Systolic blood pressure below 120 or above 145 mmHg
* Diastolic blood pressure above 95 mmHg
* Heart rate below 45 or above 95 beats / min
* Clinically relevant findings in the physical examination
* Suspicion of drug or alcohol abuse
* Regular daily consumption of more than 1 L of xanthin-containing beverages
* Intake of foods or beverages containing grapefruit within 4 weeks before the pre-study examination

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Within 48 hours after each treatment
  Maximum drug concentration in plasma after dose administration for nifedipine and candesartan
AUC(0-tn) | Within 48 hours after each treatment
  AUC from time 0 to the last data point for nifedipine and candesartan

SECONDARY OUTCOMES:
AUC | Within 48 hours after each treatment
  Area under the plasma concentration vs time curve from zero to infinity after single (first) dose for nifedipine and candesartan
Cmax,norm | Within 48 hours after each treatment
  Maximum drug concentration in plasma after dose administration divided by dose (mg) per kg body weight for nifedipine and candesartan
AUCnorm | Within 48 hours after each treatment
  Area under the curve divided by dose per kg body weight for nifedipine and candesartan
AUC(0-48) | Within 48 hours after each treatment
  AUC from time 0 to time 48 h for nifedipine and candesartan
tmax | Within 48 hours after each treatment
  Time to reach maximum drug concentration in plasma after single (first) dose for nifedipine and candesartan
t½ | Within 48 hours after each treatment
  Half-life associated with the terminal slope for nifedipine and candesartan
MRT | Within 48 hours after each treatment
  Mean residence time for nifedipine and candesartan
CL/f | Within 48 hours after each treatment
  Total body clearance of drug from plasma calculated after oral administration (apparent oral clearance) for nifedipine and candesartan
Number of participants with adverse events | Approximately 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Brendel E, Weimann B, Dietrich H, Froede C, Thomas D. Investigation of bioequivalence of a new fixed-dose combination of nifedipine and candesartan with the corresponding loose combination as well as the drug-drug interaction potential between both drugs under fasting conditions. Int J Clin Pharmacol Ther. 2013 Sep;51(9):753-62. doi: 10.5414/CP201879. PMID 23849325
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/